CLINICAL TRIAL: NCT03033888
Title: Community-Based Cervical Cancer Prevention and Education Among Women Living With HIV
Acronym: CHECC-uP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00060938; P30AI094189 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Intervention Group (Other): Intervention includes: Trained community health workers will deliver 1) 1.5-2 hour health literacy training offered in a group format at an approved community site that is most convenient to the majority of participants ; and 2) monthly phone follow-up and navigation assistance for 6 months. We will offer a Human Papilloma Virus (HPV) mobile app for participant's adolescent/young adult child (11-26 yrs), as an option rather than part of the standardized protocol. The app will be introduced at the end of the health literacy group training session for the intervention group; those who choose to download the app will be given a link with study specific password. They will be encouraged to go through the key HPV related contents with their children at home at a time that is most convenient for them.
  Interventions: Behavioral: Health-Literacy Focused Education Session
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Health-Literacy Focused Education Session
  Arms: Intervention Group

SUMMARY:
The long-term goal is to build a sustainable, community-based outreach program to promote cervical cancer screening among women living with HIV (WLH), thereby reducing related morbidity and mortality. The strategy for achieving this goal is to develop an intervention incorporating health literacy approaches and principles of community-based participatory research. Health literacy is a relatively new concept that has been applied mainly toward identifying high-risk individuals rather than toward changing health behaviors and outcomes. The proposed intervention is the first to integrate health literacy into educating WLH to promote cervical cancer screening. Community Health Workers (CHW) support has also rarely been incorporated into cancer screening interventions targeting WLH, making the proposed intervention a uniquely comprehensive approach. Building on recent successful testing by the investigators of a health literacy-focused intervention to promote cervical cancer screening in recent immigrant women, the investigators will test whether health literacy-focused interventions delivered by trained CHWs will be effective in promoting health literacy and increasing Pap test rates in a new population, WLH. The investigators hypothesize that, compared to WLH in the control group, WLH who receive the health literacy-focused CHW intervention will demonstrate: (1) higher rates of Pap test, (2) greater levels of health literacy, (3) higher levels of cervical cancer knowledge, and (4) higher self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection Able to read and write English 12+ months since Pap test Willing to provide written consent to allow the team to audit medical records for Pap test use

Exclusion Criteria:

* Had undergone a hysterectomy Pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-04; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Completion of Pap test (medical records) | 6 months
  Participants medical records will be audited to verify completion of a Pap test within 6 months of completing baseline survey. The measure of completion of Pap testing by 6 months after baseline visit will be tested using a one-sided, two-group test of proportions set at an alpha of 0.05. Known covariates of Pap test screening (e.g., age, education, insurance, and provider recommendation) will be controlled in the analyses.

SECONDARY OUTCOMES:
Change scores for health literacy | Baseline and 6 months
  Health Literacy scores will be measured using Assessment of Health Literacy-Cancer, a cervical cancer specific instrument with 52 items. Scores on the scale range from 0-52 with a score > 26 signifying a high health literacy score and scores <26 signifying low health literacy score. The rationale for using change scores is to account for differences in baseline performance for study participants, and to focus on improvement in scores after intervention. Differences in change scores between groups will be tested using a one-sided, two-group test of means with p=0.05
Change scores for cervical cancer knowledge | Baseline and 6 months
  Cervical cancer knowledge will be measured with the Cervical Cancer Knowledge Test, a 22- item which measures knowledge of cervical cancer using a binary (true/false) scale. Higher scores indicate higher cervical cancer knowledge. The rationale for using change scores is to account for differences in baseline performance for study participants, and to focus on improvement in scores after intervention. Differences in change scores between groups will be tested using a one-sided, two-group test of means with p=0.05
Change scores for self-efficacy | Baseline and 6 months
  Self-efficacy will be measured with the Self Efficacy Scale, a 4- item instrument which measures how confident a woman is in carrying out tasks in relation to Pap testing. Higher scores indicate higher self-efficacy. The rationale for using change scores is to account for differences in baseline performance for study participants, and to focus on improvement in scores after intervention. Differences in change scores between groups will be tested using a one-sided, two-group test of means with p=0.05

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No